CLINICAL TRIAL: NCT02396693
Title: Successful Extubation and Noninvasive Ventilation in Preterm Infants ≤ 1500g Terms
Brief Title: Successful Extubation and Noninvasive Ventilation in Preterm ≤ 1500g Terms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Simone Nascimento Santos Ribeiro, Phd, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUMinasGerais
Record Dates: First submitted 2015-01-28; First posted 2015-03-24 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Respiratory Distress Syndrome In Premature Infants
Keywords: Newborn; non invasive ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome In Premature Infants | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NIPPV (Experimental): NIPPV - Newborns randomized to this group underwent NIPPV, in noninvasive ventilation support intermittent, in TIME mode of the respirator.
  Interventions: Device: NIPPV
- Bubble NCPAP (Placebo Comparator): Bubble NCPAP - Newborns randomized to this group bubble NCPAP, in noninvasive ventilation continuous, in bubble NCPAP.
  Interventions: Device: Bubble NCPAP
- Ventilator NCPAP (Placebo Comparator): Ventilator NCPAP - Newborns randomized to this group ventilator NCPAP, in noninvasive ventilation continuous, in NCPAP mode of the respirator.
  Interventions: Device: Ventilator NCPAP

INTERVENTIONS:
Device: NIPPV — Ventilation with nasal intermittent positive pressure - Newborns randomized to this group underwent NIPPV, the respirators in TIME mode, set with the following settings : 5-6 centimeters of water (cmH2O) pressure positive end expiratory (PEEP); Flow rate of 6-8 liters per minute (L / min); PIP(positive inspiratory pressure) < 15 centimeters of water (cm H2O) ; respiratory frequency backup (FR) < 16 bpm; inspiratory time (IT) - 0.30 to 0.33 seconds (adjustable time constant according to the weight and baseline disease)
  Other Names: Non invasive ventilation
  Arms: NIPPV
Device: Bubble NCPAP — Bubble NCPAP - Newborns randomized to this group bubble NCPAP, adjusted with the following settings: pressure positive end expiratory (PEEP) 5-6 centimeters of water (cm H2O) and Flow 6-8 liters per minute (L / min), provided through oxygen sources and compressed air (15 liters per minute - L / min), which passes through a heated humidifier through a breathing circuit that goes to the newborn, and from him, for a plastic container (250 milliliters (ml) capacity and 14 centimeters) containing sterile distilled water, which is the bubble.
  Arms: Bubble NCPAP
Device: Ventilator NCPAP — Ventilator NCPAP - Newborns randomized to this group ventilator NCPAP, of respirators in TIME mode set with the following settings: pressure positive end expiratory (PEEP) 5-6 centimeters of water (cm H2O) and Flow 6-8 liters per minute (L / min).
  Arms: Ventilator NCPAP

SUMMARY:
Noninvasive ventilation has been used in preterm newborn with respiratory distress syndrome in an attempt to assist failure extubation. The investigators investigated failure extubation in infants gestational age less than or equal to 34 weeks and weights less than or equal to 1500 grams. Neonates were randomized to noninvasive modalities support. 101 newborns were included in this study in three groups , group 1: Nasal Intermittent Positive Pressure Ventilation (NIPPV) (n=36), group 2: Nasal Continuous Positive Airway Pressure Bubble (NCPAP bubble) (n=33) and group 3: Nasal Continuous Positive Airway Pressure Bubble Ventilator (NCPAP ventilator) (n=32)

DETAILED DESCRIPTION:
The infants were randomly allocated after extubation used a list of computer-generated randomization in NIPPV modes (with the following settings: positive inspiratory pressure (PIP) < 16 centimeters of water (cm H2O), positive end-expiratory pressure (PEEP) 4-5 centimeters of water (cm H2O, backup respiratory rate (RR) < 18 cycles per minute flow 6-7 liters per minute (L / min) and inspiratory time (TI) according to the time constant for idae (0.30 to 0.34 seconds), and respirator seal to NCPAP water tower was adjusted to 4-5 centimeters of water (cm H2O) PEEP, flow 6-7 liters per minute (L / Min.) oxygen for both was adjusted to maintain arterial oxygen saturation between 85-95%

The criteria for extubation were defined using a protocol by the clinic staff, confirmed by arterial blood gases and chest X-ray, as well as adjustments of the ventilator settings.

Vital signs, blood gas parameters and noninvasive brackets were recorded before, immediately, 15, 30, 45 minutes, 1(hour) h, 2h, 12h, 24h and 48 h after extubation were documented.

Neonatal morbidities were documented until discharge, among these are: patent ductus arterious, necrotizing enterocolitis, retinopathy of prematurity, intracranial hemorrhage and pneumothorax.

Data on achievement of prenatal, antenatal steroids and surfactant administration were documented. All newborns were natural porcine surfactant Curosurf®.

The total duration of mechanical ventilation and oxygen were documented from birth until discharge or death. The supplemental oxygen or mechanical ventilation days was defined as daily requirement of fraction of inspired oxygen (FiO 2)> 0.21 or ventilation > 12 hours, respectively.

The newborns were followed for all interaction until discharge (about 5 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Were eligible for the study
* Newborn (NB) ≤ 34 weeks and 500g to the weight of ≤ 1500 grams with a diagnosis of respiratory distress syndrome (RDS) who had their first elective extubation.

Exclusion Criteria:

* Excluded patients with cardiorespiratory system malformations
* Genetic disorders
* Neuromuscular disease and malformations of the central nervous system.

Ages: 26 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2012-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The success rate of the extubation | Finished The newborns were followed for all interaction until discharge (about 5 weeks).
  The success rate of the extubation and Need for intubation within the first 48 hours after extubation in the three groups

SECONDARY OUTCOMES:
Correlations of the noninvasive support (correlations with sex, gestational age (IG), total duration of oxygen use, full-time use of mechanical ventilation and bronchopulmonary dysplasia (DBP) | Finished The newborns were followed for all interaction until discharge (about 5 weeks).
  Related to noninvasive support and correlations with sex, gestational age (IG), total duration of oxygen use, full-time use of mechanical ventilation and bronchopulmonary dysplasia (DBP).
The failure and success of the noninvasive support (days of oxygen use, mechanical ventilation (VPM) and occurrence of bronchopulmonary dysplasia (BPD) | Finished The newborns were followed for all interaction until discharge (about 5 weeks).
  The failure vs. success, with the days of oxygen use, mechanical ventilation (VPM) and occurrence of bronchopulmonary dysplasia (BPD)
Incidence of the diseases during the hospitalization | Finished The newborns were followed for all interaction until discharge (about 5 weeks).
  Incidence of pneumothorax, patent ductus arterious (PDA), retinopathy of prematurity (HOP), peri-intraventricular hemorrhage (HPIV), bronchopulmonary dysplasia (BPD), necrotizing enterocolitis (NEC), nasal injury
Outcomes at discharge in days (Total number of days in use oxygen, mechanical ventilation and death, and hospitalization duration) | Finished The newborns were followed for all interaction until discharge (about 5 weeks).
  Total number of days in use oxygen, mechanical ventilation and death, and hospitalization duration

CONTACTS AND LOCATIONS:
Overall Officials: Cíntia Johnston, Study Chair — Federal University of São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jasani B, Nanavati R, Kabra N, Rajdeo S, Bhandari V. Comparison of non-synchronized nasal intermittent positive pressure ventilation versus nasal continuous positive airway pressure as post-extubation respiratory support in preterm infants with respiratory distress syndrome: a randomized controlled trial. J Matern Fetal Neonatal Med. 2016;29(10):1546-51. doi: 10.3109/14767058.2015.1059809. Epub 2015 Jul 28. PMID 26135774
- [Result] Mehta P, Berger J, Bucholz E, Bhandari V. Factors affecting nasal intermittent positive pressure ventilation failure and impact on bronchopulmonary dysplasia in neonates. J Perinatol. 2014 Oct;34(10):754-60. doi: 10.1038/jp.2014.100. Epub 2014 May 29. PMID 24875408
- [Result] Bhandari V. Noninvasive respiratory support in the preterm infant. Clin Perinatol. 2012 Sep;39(3):497-511. doi: 10.1016/j.clp.2012.06.008. PMID 22954265
- [Result] Meneses J, Bhandari V, Alves JG. Nasal intermittent positive-pressure ventilation vs nasal continuous positive airway pressure for preterm infants with respiratory distress syndrome: a systematic review and meta-analysis. Arch Pediatr Adolesc Med. 2012 Apr;166(4):372-6. doi: 10.1001/archpediatrics.2011.1142. PMID 22474063
- [Result] Kirpalani H, Millar D, Lemyre B, Yoder BA, Chiu A, Roberts RS; NIPPV Study Group. A trial comparing noninvasive ventilation strategies in preterm infants. N Engl J Med. 2013 Aug 15;369(7):611-20. doi: 10.1056/NEJMoa1214533. PMID 23944299
- [Result] Khorana M, Paradeevisut H, Sangtawesin V, Kanjanapatanakul W, Chotigeat U, Ayutthaya JK. A randomized trial of non-synchronized Nasopharyngeal Intermittent Mandatory Ventilation (nsNIMV) vs. Nasal Continuous Positive Airway Pressure (NCPAP) in the prevention of extubation failure in pre-term < 1,500 grams. J Med Assoc Thai. 2008 Oct;91 Suppl 3:S136-42. PMID 19253509
- [Result] Bahman-Bijari B, Malekiyan A, Niknafs P, Baneshi MR. Bubble-CPAP vs. Ventilatory-CPAP in Preterm Infants with Respiratory Distress. Iran J Pediatr. 2011 Jun;21(2):151-8. PMID 23056781
- [Result] Kumar M, Avasthi S, Ahuja S, Malik GK, Singh SN. Unsynchronized Nasal Intermittent Positive Pressure Ventilation to prevent extubation failure in neonates: a randomized controlled trial. Indian J Pediatr. 2011 Jul;78(7):801-6. doi: 10.1007/s12098-010-0357-x. Epub 2011 Feb 2. PMID 21287368